CLINICAL TRIAL: NCT06227143
Title: Monitoring Depth of Anesthesia During Opioid Free Anesthesia
Brief Title: Anesthesia Depth During Opioid Free Anesthesia
Status: Completed | Type: Observational
Sponsor: Region Halland (Other)
Responsible Party: Principal Investigator, Anna Persson, MD, PhD, Consultant in Anaesthesia and Intensive Care Medicine, Region Halland
Other Study IDs: 2022-07156-02
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Opioid-free Anesthesia; Anesthesia Depth Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Opioid-free anesthesia: Patients undergoing laparoscopic surgery under general anesthesia. Drugs used for the purpose of anesthesia:
  Ketamine Dexmedetomidine Propofol Sevoflurane Lidocaine Betamethasone Paracetamol NSAID
  Interventions: Procedure: Anesthesia depth monitoring
- Target Controlled Infusion: Patients undergoing laparoscopic surgery under general anesthesia. Drugs used for the purpose of anesthesia:
  Propofol Remifentanil Oxycodone Paracetamol NSAID Bethametasone
  Interventions: Procedure: Anesthesia depth monitoring
- Volatile anesthetics: Patients undergoing laparoscopic surgery under general anesthesia. Drugs used for the purpose of anesthesia:
  Sevoflurane Propofol Remifentanil Oxycodone Paracetmol NSAID Bethametasone
  Interventions: Procedure: Anesthesia depth monitoring

INTERVENTIONS:
Procedure: Anesthesia depth monitoring — Anesthesia depth monitoring during opioid-free anesthesia

SUMMARY:
Opioid-free anesthesia is feasible and effective but still not common practice. Anesthesia depth monitoring is not investigated for use in anesthesia combining low dose infusions of several drugs with different sedative patterns on EEG. This is an observational study comparing opioid-free anesthesia with regular anesthesia in regards to DSA, SEF and PSI from the Sedline monitor.

DETAILED DESCRIPTION:
Patients who undergo general anaesthesia are more or less extensively monitored, with the sole purpose of surveilling depth of anesthesia and nociception. Parameters such as heart rate, blood pressure, pupillary size and sweating has historically been used as predictive markers for this surveillance. However, these clinical parameters have low predictive capacity and there is a tendency to overdue perioperative sedation and misinterpret sympathetically derived reactions as pain. This could lead to higher incidence of postoperative delirium and opioid induced hyperalgesia. On the contrary, an overestimated trust in the mentioned parameters might lead to increased risk of intra-operative awareness.

The usefulness of processed encephalography (pEEG) during anesthesia has since long been promoted for anesthesia providers. Since then, several commercial devices has been developed and deployed for clinical use. Although mixed results are presented in clinical studies there is now a significant empirical experience for its use in routine anesthesia with volatile anesthetics and propofol. Density spectral array (DSA) is the latest contribution in the field of encephalographic monitoring. It is a two-dimensional graph plotting the power of each frequency-interval on a time-scale.

More and more data on the effectiveness and safety of opioid free anaesthesia (OFA) have been released, especially as a direct result of the ongoing opioid-epidemic affecting a large number of people worldwide. The algorithms for the commercial devices, using DSA, has to this date not been validated for multimodal anesthetic regimens using ketamine and dexmedetomidine.

The purpose of this observational study is to compare DSA pattern and data for pEEG between OFA and total intravenous anaesthesia or general anaesthesia with volatile anesthetics for patients undergoing laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic surgery
* Adult patients
* Ability to accomodate verbal and written information in swedish
* Voluntary

Exclusion Criteria:

* Pregnancy
* Intolerance to NSAID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing laparoscopic surgery under general anesthesia with different protocol-based anesthetic methods (opioid-free, intravenous target controlled or volatile) included after written and oral consent.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Patient state index level (PSI) | 20 minute during steady state peroperative anesthesia
  Difference in PSI levels during opioid-free anesthesia, target controlled and volatile anesthesia measured with Kruskal-Wallis

SECONDARY OUTCOMES:
Spectral edge frequency (SEF) | 20 minute during steady state peroperative anesthesia
  Difference in SEF levels during opioid-free anesthesia, target controlled and volatile anesthesia measured with Kruskal-Wallis

OTHER OUTCOMES:
Density Spectral Array (DSA) | 20 minute during steady state peroperative anesthesia
  Descriptive comparison of DSA appearance during opioid-free anesthesia, target controlled and volatile anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Krister Mogianos, MD, Principal Investigator — Region Halland
Locations (1):
- Halland Hospital Halmstad, Halmstad, Halland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Project plan. Individual measurements. Statistical analysis.

REFERENCES:
- [Derived] Mogianos K, Persson AK. Anesthesia depth monitoring during opioid free anesthesia - a prospective observational study. BMC Anesthesiol. 2025 Jan 24;25(1):37. doi: 10.1186/s12871-024-02859-1. PMID 39856547